CLINICAL TRIAL: NCT00652717
Title: A Multicenter, Open Study To Evaluate The Efficacy Of Ezetimibe 10 Mg Added On Statin Therapy, In Reducing LDL Cholesterol To Target Levels In Patients After Acute Coronary Syndrome
Brief Title: Study To Assess The Efficacy Of A Cholesterol Lowering Drug On Top Of Statins In Patients After Myocardial Infarction (MI)(0653A-150)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-150; 2008_009
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Disorder
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ezetimibe; Simvastatin

ARMS (2):
- 1 (Experimental): arm 1 - Ezetimibe 10 mg daily that was added on Statin Therapy (prescribed clinically suitable dose by the physician).
  Interventions: Drug: Ezetimibe; Drug: simvastatin
- 2 (Active Comparator): arm 2- simvastatin (prescribed clinically suitable dose by the physician), for mean follow up of 42 days.
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 10 mg daily for 42 days.
  Other Names: Ezetrol®; Zetia®; MK0653
  Arms: 1
Drug: simvastatin — simvastatin (prescribed clinically suitable dose by the physician), for mean follow up of 42 days.
  Other Names: Zocor®; MK0733

SUMMARY:
Collecting local data, safety and experience trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients; Post Acute Coronary Syndrome

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2005-02-01 (Actual); Primary Completion 2005-02-15 (Actual); Study Completion 2005-08-04 (Actual)

PRIMARY OUTCOMES:
LDL levels | 42 Days

SECONDARY OUTCOMES:
Safety measures | 42 days
Total cholesterol levels. | 42 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC